CLINICAL TRIAL: NCT02016300
Title: Effects of Unloader Bracing in Clinical Outcome and Articular Cartilage Physiology Following Microfracture of Isolated Chondral Defects
Brief Title: Effects of Unloader Bracing in Clinical Outcome and Cartilage Physiology Following Microfracture of Chondral Defects
Acronym: Mfxbracing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jason L. Dragoo, Associate Professor of Orthopaedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: oss-mfx-2013
Record Dates: First submitted 2013-12-02; First posted 2013-12-19 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-05

CONDITIONS: Cartilage Loss; Microfracture
Keywords: cartilage; microfracture; knee; bracing
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unloader Bracing (Experimental): This group will be randomly selected and assigned to wear an unloader brace post-operatively during the study period.
  Interventions: Device: Unloader Bracing
- Non-Bracing Arm (Active Comparator): This group will be randomly selected and assigned to wear no brace post-operatively.
  Interventions: Device: Non-Bracing

INTERVENTIONS:
Device: Unloader Bracing — The bracing arm patients will be randomly selected and will wear an unloader brace post-operatively during the study period.
  Other Names: Ossur Unloader Brace
  Arms: Unloader Bracing
Device: Non-Bracing — Microfracture performed with no post-operative unloader bracing
  Arms: Non-Bracing Arm

SUMMARY:
The study will examine clinical and radiographic outcomes of microfracture surgery (a common technique to address isolated areas of cartilage loss) in the knee used with or without unloader bracing. Randomly selected patients will wear an unloader brace, which is designed to take pressure off the area of the knee which underwent repair, for several weeks after surgery. Our hypothesis is that bracing may improve clinical and or radiographic outcomes.

The surgery performed will be the same for all patients

The length of follow up and schedule of post-operative MRI will be the same for all patients.

The only difference in groups will be presence of absence of brace wear.

DETAILED DESCRIPTION:
The study will examine clinical and radiographic outcomes of microfracture surgery (a common technique to address isolated areas of cartilage loss) in the knee used with or without unloader bracing. Radiographic outcome will be assessed via MRI scans post-operatively. Randomly selected patients will wear an unloader brace, which is designed to take pressure off the area of the knee which underwent repair, for several weeks after surgery. Our hypothesis is that bracing may improve clinical and or radiographic outcomes.

The surgery performed will be the same for all patients

The length of follow up and schedule of post-operative MRI will be the same for all patients.

The only difference in groups will be presence of absence of brace wear.

ELIGIBILITY:
Inclusion Criteria:

* isolated chondral defect of medial or lateral femoral condyle 2cm squared or less
* age 15-40
* neutral knee alignment

Exclusion Criteria:

* prior cartilage procedures performed in the same knee
* other significant knee pathology including meniscus tears, ligament tears or inflammatory arthritis

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Dragoo, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Unloader Bracing: This group was randomly selected and assigned to wear an unloader brace post-operatively during the study period.
- Non-Bracing Arm: This group was randomly selected and assigned to wear no brace post-operatively.
Period: Overall Study
Arm/Group | Unloader Bracing | Non-Bracing Arm
Started | 12 | 12
Completed | 12 | 9
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Unloader Bracing | Non-Bracing Arm | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (8.5) | 39.6 (10.2) | 40.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 9 | 21
  Unknown or Not Reported | 0 | 0 | 0
Knee Injury and Osteoarthritis Outcome Score (KOOS) [Mean (Standard Deviation); unit: units on a scale] — Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
  units on a scale | 76.8 (18.9) | 79.6 (16.1) | 78.0 (17.4)
Tegner Score [Mean (Standard Deviation); unit: units on a scale] — The Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity and that before injury. A score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports. A score >6 can only be achieved if the person participates in recreational or competitive sport.
  units on a scale | 2.2 (1.3) | 2.0 (1.9) | 2.1 (1.6)
SF-12 Score [Mean (Standard Deviation); unit: units on a scale] — SF-12 scale is a generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey which, when combined, scored and weighted, results in two scales of mental and physical functioning and overall health-related quality of life. A higher value indicates a better quality of life of the patient. The scores range from 0 to 100.
  units on a scale | 28.8 (2.9) | 28.9 (2.4) | 28.8 (2.6)
Lysholm Score [Mean (Standard Deviation); unit: units on a scale] — The Lysholm score is an indexed score of knee functional ability, with 0 being the worst score and 100 being the best score, indicating no limitations in activity/function.
  units on a scale | 63.6 (24.7) | 51.3 (24.7) | 58.3 (24.9)
T2 Relaxation time [Mean (Standard Deviation); unit: milliseconds (ms)] — T2 imaging assesses hydration of cartilage as well as collagen fiber orientation and loss of type II collagen.
  milliseconds (ms) | 31.4 (38.1) | 42.8 (96.8) | 36.5 (68.3)
Cartilage Volume [Mean (Standard Deviation); unit: mm^3] — Negative values indicate that the reading was less than the reference zone for cartilage volume.
  mm^3 | -6.5 (36.3) | -6.3 (46.3) | -6.4 (39.8)
Cartilage Thickness [Mean (Standard Deviation); unit: mm] — Negative values indicate that the reading was less than the reference zone for cartilage thickness.
  mm | -0.1 (0.3) | -0.2 (0.4) | -0.1 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) (Clinical Outcome)
Description: KOOS is a validated outcome score that evaluates knee symptoms, knee pain, knee use in activities of daily living, function in sport and recreation and knee-related quality of life. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Time Frame: 2 years
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unloader Bracing | Non-Bracing Arm
Number analyzed (Participants) | 12 | 9
units on a scale
  Change at month 6 | 12.0 (12.2) | 4.1 (12.2)
  Change at month 12 | 19.1 (16.9) | 8.1 (11.5)
  Change at month 24 | 17.8 (16.7) | 4.6 (10.3)
Statistical Analysis 1: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 6; Test type: Other; p = 0.162, Regression, Linear
Statistical Analysis 2: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 12; Test type: Other; p = 0.094, Regression, Linear
Statistical Analysis 3: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 24; Test type: Other; p = 0.043, Regression, Linear

2. Secondary Outcome: Change From Baseline in Tegner Score (Clinical Outcome)
Description: The Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity and that before injury. A score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports. A score >6 can only be achieved if the person participates in recreational or competitive sport.
Time Frame: 2 years
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unloader Bracing | Non-Bracing Arm
Number analyzed (Participants) | 12 | 9
units on a scale
  Change at month 6 | 1.7 (1.2) | 0.9 (2.6)
  Change at month 12 | 2.7 (1.1) | 1.9 (2.2)
  Change at month 24 | 2.3 (1.9) | 1.4 (1.2)
Statistical Analysis 1: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 6; Test type: Other; p = 0.387, Regression, Linear
Statistical Analysis 2: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 12; Test type: Other; p = 0.340, Regression, Linear
Statistical Analysis 3: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 24; Test type: Other; p = 0.179, Regression, Linear

3. Secondary Outcome: Change From Baseline in SF-12 Quality of Life Score (Clinical Outcome)
Description: SF-12 scale is a generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey which, when combined, scored and weighted, results in two scales of mental and physical functioning and overall health-related quality of life. A higher value indicates a better quality of life of the patient. The scores range from 0 to 100.
Time Frame: 2 years
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unloader Bracing | Non-Bracing Arm
Number analyzed (Participants) | 12 | 9
units on a scale
  Change at month 6 | 2.2 (3.0) | 2.9 (5.5)
  Change at month 12 | 2.4 (4.1) | 2.3 (3.0)
  Change at month 24 | 0.8 (5.1) | 2.1 (6.8)
Statistical Analysis 1: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 6; Test type: Other; p = 0.729, Regression, Linear
Statistical Analysis 2: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 12; Test type: Other; p = 0.958, Regression, Linear
Statistical Analysis 3: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 24; Test type: Other; p = 0.634, Regression, Linear

4. Secondary Outcome: Change From Baseline in Lysholm Score (Clinical Outcome)
Description: The Lysholm score is an indexed score of knee functional ability, with 0 being the worst score and 100 being the best score, indicating no limitations in activity/function.
Time Frame: 2 years
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unloader Bracing | Non-Bracing Arm
Number analyzed (Participants) | 12 | 9
units on a scale
  Change at month 6 | 14.3 (16.2) | 11.1 (23.1)
  Change at month 12 | 25.7 (33.9) | 20.3 (21.7)
  Change at month 24 | 20.3 (20.5) | 18.8 (17.1)
Statistical Analysis 1: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 6; Test type: Other; p = 0.733, Regression, Linear
Statistical Analysis 2: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 12; Test type: Other; p = 0.666, Regression, Linear
Statistical Analysis 3: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 24; Test type: Other; p = 0.854, Regression, Linear

5. Secondary Outcome: Change From Baseline in T2 Relaxation Time (Radiographic Outcome)
Description: T2 imaging assesses hydration of cartilage as well as collagen fiber orientation and loss of type II collagen.
Time Frame: 2 years
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Unloader Bracing | Non-Bracing Arm
Number analyzed (Participants) | 12 | 9
millisecond (ms)
  Change at month 12 | -24.5 (25.3) | -36.2 (73.8)
  Change at month 24 | -25.1 (25.1) | -17.6 (5.6)
Statistical Analysis 1: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 12; Test type: Other; p = 0.774, Regression, Linear
Statistical Analysis 2: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 24; Test type: Other; p = 0.414, Regression, Linear

6. Secondary Outcome: Change From Baseline in Cartilage Volume (Radiographic Outcome)
Time Frame: 2 years
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Unloader Bracing | Non-Bracing Arm
Number analyzed (Participants) | 12 | 9
mm^3
  Change at month 12 | 31.4 (31.8) | -2.1 (37.5)
  Change at month 24 | 49.2 (35.8) | 17.8 (52.3)
Statistical Analysis 1: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 12; Test type: Other; p = 0.064, Regression, Linear
Statistical Analysis 2: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 24; Test type: Other; p = 0.276, Regression, Linear

7. Secondary Outcome: Change From Baseline in Cartilage Thickness (Radiographic Outcome)
Time Frame: 2 years
Population: Participants who completed the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Unloader Bracing | Non-Bracing Arm
Number analyzed (Participants) | 12 | 9
mm
  Change at month 12 | 0.3 (0.3) | -0.2 (0.4)
  Change at month 24 | 0.3 (0.3) | 0.1 (0.2)
Statistical Analysis 1: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 12; Test type: Other; p = 0.020, Regression, Linear
Statistical Analysis 2: Comparison: Unloader Bracing vs Non-Bracing Arm; Difference between baseline and month 24; Test type: Other; p = 0.091, Regression, Linear

ADVERSE EVENTS:
Time Frame: Up to two years.
Arm/Group | Unloader Bracing | Non-Bracing Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2011-12-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT02016300/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT02016300/SAP_001.pdf